CLINICAL TRIAL: NCT02653586
Title: "In Favor of Resilience Self" Prevention Program Promoting Positive Self-Image and Body Image Among Adolescence Aged 15-17
Brief Title: Prevention Program Promoting Self Resilience,Positive Self-Image and Body Image Among Adolescence Aged 15-17
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Hai College (Other)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, shani aboutboul, principal investigator, Tel Hai College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: telhaicolege
Record Dates: First submitted 2016-01-03; First posted 2016-01-12 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Primary Prevention
Keywords: resilience; prevention program; body image; self esteem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- program "In Favor of Resilience Self" (Experimental): The program "In Favor of Resilience Self" was delivered to adolescence aged 15-17, over 2 months. The program contained nine weekly, 90-min lessons that focus on enhancing self- resilience, self-esteem, self-image, body image. All students completed a self-report questionnaire at baseline, conclusion and 3 months after program conclusion.
  Interventions: Other: program "In Favor of Resilience Self"
- control group (No Intervention): The control group didn't receive the intervention program, instead they received a lecture on wised nutrition. In addition the control group completed the same self-report questionnaire as the intervention group at baseline, conclusion and 3 months after program.

INTERVENTIONS:
Other: program "In Favor of Resilience Self" — A prevention program aiming at improve self-resilience ,self-esteem and body image, contains nine interactive activities, based on a cognitive dissonance method.
  Other Names: "In Favor of myself"
  Arms: program "In Favor of Resilience Self"

SUMMARY:
The study was a group randomized controlled trial. Within each school Classes of high school students were allocated by randomization to the intervention or control group by a function Randomization in Excel program. Outcomes were measured by questionnaire at pre- intervention, post-intervention and 3-month follow-up. The study protocol was approved by Tel Hai college institutional review board. Parents of all participants, in the intervention and in the control group, received information about the program and the study and were choose whether to provided informed consent or not.

DETAILED DESCRIPTION:
Participants and setting Two high schools were recruited for the study, in each school classes from grades 9th and 10th were chosen to participate in the study all mixed gender classes. The two high schools are in northern Israel, one in a rural area and the second in a small city, both serving the Jewish population. The size of the schools were similar. All data were collected within the school setting.

Program description "Towards a more resilient self" is an interactive, cognitive behavior program aiming to address low resilience, low self-esteem and body dissatisfaction. The program contains a range of coping strategies to help adolescents improve resilience, self-esteem and body image. The program consists of nine 90-min sessions delivered by one group leader in the presence of the classes' teachers. Participants in the control group received one session of 90 minutes with health nutrition education.

ELIGIBILITY:
Inclusion Criteria:

* Participants who filled out the questionnaires before and after the program, and if their parents have signed a letter of agreement

Exclusion Criteria:

* Participants who do not completed the questionnaires at least twice

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 209 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The Connor-Davidson Resilience Scale (CD-RISC) | Measured three times during six months, measuring a change in resilience scale
  The CD-RISC contains 25 items, all of which carry a 5-point range of responses, as follows: not true at all (0), rarely true (1), sometimes true (2), often true (3), and true nearly all of the time (4). The scale is rated based on how the subject has felt over the past month. The total score ranges from 0-100, with higher scores reflecting greater resilience. Examples of questions: "Able to adapt to change", "Think of self as strong person"
Rosenberg self esteem scale | Measured three times during six months, measuring a change in rosenberg self esteem scale
  The scale is a ten item Likert scale with items answered on a four point scale - from strongly agree- (3), agree (2), disagree (1), strongly disagree (0). The total score ranges from 0-30 The higher the score, the higher the self esteem.
  to strongly disagree.

REFERENCES:
- [Derived] Agam-Bitton R, Abu Ahmad W, Golan M. Girls-only vs. mixed-gender groups in the delivery of a universal wellness programme among adolescents: A cluster-randomized controlled trial. PLoS One. 2018 Jun 18;13(6):e0198872. doi: 10.1371/journal.pone.0198872. eCollection 2018. PMID 29912918